CLINICAL TRIAL: NCT01201447
Title: Prevalence of Questionable Occlusal Caries Lesions
Brief Title: DPBRN Prevalence of Questionable Occlusal Caries Lesions
Status: Completed | Type: Observational
Sponsor: Dental Practice-Based Research Network (Network)
Collaborators: HealthPartners Institute (Other); Kaiser Permanente (Other); Permanente Dental Associates Group, Oregon (Other); National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Gregg H. Gilbert, DDS MBA, Study Chair, University of Alabama at Birmingahm
Other Study IDs: 119275; U01DE016747 (NIH)
Record Dates: First submitted 2010-09-13; First posted 2010-09-14 (Estimated); Last update posted 2011-03-04 (Estimated); Status verified 2011-03

CONDITIONS: Dental Caries
Keywords: Assessment; Questionable Caries
MeSH Terms: conditions — Dental Caries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Questionable occlusal lesions

SUMMARY:
The purpose of this study was to investigate the process involved when making decisions about the diagnosis and treatment of questionable lesions, as well as determine if there is any association between lesions progression (or depth, if opened) and clinical characteristics and baseline risk assessment.

DETAILED DESCRIPTION:
The term"questionable" is defined as a tooth with no cavitation (no continuity break in the enamel) and no radiographic radiolucencies, but the presence of caries is suspected due to roughness, surface opacities, or staining. The characteristics of these lesions and the patient's baseline caries risk were examined.

There have been very few studies regarding questionable lesions, virtually no clinical evaluations of the progression of questionable lesions over time, and no studies depicting the prevalence of these lesions. Since carious lesions have the ability to arrest and possibly reverse, determining how often these lesions are being seen in practice and learning more about their characteristics and patient risk assessment are important steps in order to manage these lesions without unnecessary surgical intervention.

ELIGIBILITY:
Inclusion Criteria:

* patients needed to have at least one permanent tooth with a questionable lesion. This means that subjects were at least 6 years old because that is when the permanent first molar typically erupts.

Exclusion Criteria:

* patients under 6 years old
* patients 6 years old and older who do not have a questionable lesion

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The participants directly involved in this study were the patients who have sought dental treatment in the DPBRN practitioner-investigators' practices.
Sampling Method: Non-Probability Sample
Enrollment: 2624 (Estimated)
Dates: Start 2008-08; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonia K Makhija, DDS, MPH, Principal Investigator — University of Alabama at Birmingham
Locations (7):
- United States (6):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of Florida College of Dentistry, Gainesville, Florida
  - Health Partners Dental Group, Minneapolis, Minnesota
  - Health Partners Research Foundation, Minneapolis, Minnesota
  - Kaiser Permanente Center for Health Research, Portland, Oregon
  - Permanente Denrtal Associates, Portland, Oregon
- University of Copenhagen Royal Dental College, Copenhagen, Denmark

REFERENCES:
- See also: Dental Practice-Based Research Network — http://DPBRN.org
- See also: Dental Practice-Based Research Network — http://DentalPBRN.org